CLINICAL TRIAL: NCT01384331
Title: Phase 4 Study Comparison of Two Combined Oral Contraceptive Regimens and an Intravaginal Hormonal Ring Against Placebo for Management of Bleeding Problems in Women Using Implanon, the Sub-dermal Contraceptive Implant
Brief Title: New Treatments for Troublesome Bleeding in Implanon Users
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Family Planning Association New South Wales (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Edith Weisberg, Sydney Centre for Reproductive Health Research, Family Planning NSW
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2011-01; ACTRN12611000617965 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Menstrual Problem
Keywords: Implanon users; Frequent bleeding; Prolonged bleeding; Comparison of treatments; Placebo controlled; Randomly allocated tretment
MeSH Terms: conditions — Menstruation Disturbances | interventions — Desogestrel; NuvaRing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 Marvelon ,placebo (Active Comparator): 7 days daily intake of oral capsule containing "Marvelon" ethinyl oestradiol 30micrograms plus desogestrel 150 micrograms followed by 14 days oral placebo capsules containing starch for 21 day treatment Cycle
  Interventions: Drug: Marvelon
- Marvelon (Active Comparator): * 21 days daily intake of oral capsules containing ethinyl oestradiol 30micrograms plus desogestrel 150 micrograms
  * for one cycle of 21 days
  Interventions: Drug: Marvelon
- NuvaRing (Active Comparator): 21 days NuvaRing contraceptive vaginal ring releasing ethinyl oestradiol 15micrograms plus etonorgestrel 120 micrograms dailyleft in situ for 21 days Treatment will be for 21 days
  Interventions: Drug: Marvelon
- Starch capsule (Placebo Comparator): 21 days daily oral placebo capsules Treatment will be for one 21 day cycle
  Interventions: Drug: Marvelon

INTERVENTIONS:
Drug: Marvelon — 7 days daily intake of oral capsule containing containing ethinyl oestradiol 30micrograms plus desogestrel 150 micrograms followed by 14 days oral placebo capsules
  * 21 days daily intake of oral capsules containing ethinyl oestradiol 30micrograms plus desogestrel 150 micrograms
  * 21 days NuvaRing contraceptive vaginal ring releasing ethinyl oestradiol 15micrograms plus etonorgestrel 120 micrograms dailyleft in situ for 21 days
  * 21 days daily oral placebo capsules Treatment will be for one cycle of 21 days
  Other Names: NuvaRing

SUMMARY:
Most Implanon users experience a reduction in the frequency and volume of menstrual bleeding, but a substantial minority experience unpredictable and frequent and/or prolonged episodes of bleeding. This is a double blind, placebo controlled, randomised study with an additional randomised non-blinded arm. Two hundred women between the ages of 18-45 years, who are Implanon users with prolonged or frequent breakthrough bleeding (WHO definition) will be recruited and randomised into 4 equal-sized treatment groups of 50 women assigned to Marvelon 7 days or 21 days, NuvaRing 21 days or placebo. Recruited subjects will maintain a daily menstrual diary chart for a minimum of 90 days prior to randomisation, and will be enrolled into the treatment phase provided that they have met one of the World Health Organization criteria for prolonged or frequent bleeding Following the initial 90 day record, eligible women will begin designated treatment on day 1 of the next episode of bleeding or spotting. Analysis of the subsequent menstrual pattern will begin from day 1 of that bleeding/spotting episode and will continue through 90 days.

DETAILED DESCRIPTION:
This is a double blind, placebo controlled, randomised study with an additional randomised non-blinded arm. Two hundred women between the ages of 18-45 years, who are Implanon users with prolonged or frequent breakthrough bleeding (WHO definition) will be recruited and randomised into 4 equal-sized treatment groups of 50 women assigned to Marvelon 7 days or 21 days, NuvaRing 21 days or placebo. Recruited subjects will maintain a daily menstrual diary chart for a minimum of 90 days prior to randomisation, and will be enrolled into the treatment phase provided that they have met one of the World Health Organization criteria for prolonged or frequent bleeding (in the 90 day reference period one episode of bleeding and/or spotting lasting > 10 days, or more than 4 bleeding/spotting episodes). Randomisation will be performed by computer generation of a random number table in blocks of ten, with equal numbers in each of the four groups. The medications will be packed in sequentially numbered and sealed opaque envelopes (independent of the investigators).

Following the initial 90 day record, eligible women will begin designated treatment on day 1 of the next episode of bleeding or spotting. Analysis of the subsequent menstrual pattern will begin from day 1 of that bleeding/spotting episode and will continue through 90 days. Analysis of the pre-treatment menstrual pattern will include the 90 days immediately preceding the bleeding episode in which treatment starts.

Women will participate in the study for approximately seven months depending on their bleeding pattern.

Data analysis:

Data will be analysed on an intention to treat basis, entered on SPSS and analysed prior to breaking the randomisation code. Frequency analyses will be undertaken for demographic data and means (SD) compared to check effectiveness of the randomisation scheme. Total number of days of spotting, bleeding, bleeding and spotting and number of episodes during the pre and post 90 days reference period will be entered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-45 using the subdermal progestogen-only contraceptive implant and experiencing frequent or prolonged vaginal bleeding Willing to keep a menstrual diary for 6 months

Exclusion Criteria:

Women who have currently or previously had

* Heart attack or stroke
* Blood clot in a vein
* High blood pressure
* Severe liver or kidney disease
* Blood pressure > 135 mm systolic or >85 mm diastolic
* Migraine with aura
* Breast cancer or any genital cancer
* Severe chronic liver or kidney disease
* Women with known sensitivity to ethinyl oestradiol, progestogens
* Women taking phenytoin, carbamazepine or phenobarbitol
* Women who are pregnant
* Women who are lactating
* Women who are unwilling to keep a daily menstrual diary or otherwise unwilling to follow the study criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The number of days to stop bleeding after initiation of each treatment group and placebo | Within 3 weeks of starting therapy
  The number of days to stop bleeding after initiation of each treatment group and placebo determined from menstrual diaries completed by subjects

SECONDARY OUTCOMES:
The mean total number of bleeding and spotting days during the 90 day "treatment" reference period | Six months after entering study
  The mean total number of bleeding and spotting days during the 90 day "treatment" reference period compared with the pre-treatment reference period (calculated as percentage reduction) for each group and a comparison between treatment groups and placebo and compared to the other treatment groups determined from menstrual diaries kept for 90 days prior to starting treatment and for 90 days from initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Weisberg, MB BS MM, Principal Investigator — Family Planning NSW; Ian S FRASER, BSC MD, Principal Investigator — University of Sydney
Locations (1):
- Sydney centre for Reproductive Health Research, FPNSW, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Weisberg E, Hickey M, Palmer D, O'Connor V, Salamonsen LA, Findlay JK, Fraser IS. A randomized controlled trial of treatment options for troublesome uterine bleeding in Implanon users. Hum Reprod. 2009 Aug;24(8):1852-61. doi: 10.1093/humrep/dep081. Epub 2009 Apr 15. PMID 19369294